CLINICAL TRIAL: NCT03222089
Title: FOLFOXIRI in Combination With GM-CSF and IL-2 (FOLFOXIGIL) Versus FOLFOXIRI as First-line Treatment for Patients With Metastatic Colorectal Cancer: a Phase II Trial by the FNF Team.
Brief Title: Phase II Trial of FOLFOXIGIL Versus FOLFOXIRI as First-line Therapy in Patients With mCRC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Another study enrolling the similar group of patient are ongoing
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNF-006
Record Dates: First submitted 2017-07-03; First posted 2017-07-19 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Oxaliplatin; Levoleucovorin; Fluorouracil; Granulocyte-Macrophage Colony-Stimulating Factor; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFOXIGIL (Experimental): The FOLFOXIGIL chemoimmunotherapy regimen is composed by FOLFOXIRI chemotherapy and the immunotherapy of GM-CSF and IL-2.
  FOLFOXIRI: Irinotecan 165 mg/m² + oxaliplatin 85 mg/m² + Levoleucovorin 200 mg/m² + 5-FU 2800 mg/m² cont. inf. 46h all on day 1, repeated every 2 weeks.
  GM-CSF 150ug s.c. d3-7; Interleukin-2 100MIU s.c. d8-14 and d17-d28, Repeated every 4 weeks.
  Treatment will be administered until progression, patients' withdrawal of consent, unacceptable toxicity.
  Interventions: Drug: Irinotecan; Drug: Oxaliplatin; Drug: Levoleucovorin; Drug: 5-FU; Drug: GM-CSF; Drug: IL-2
- FOLFOXIRI (Active Comparator): Irinotecan 165 mg/m² + oxaliplatin 85 mg/m² + Levoleucovorin 200 mg/m² + 5-FU 2800 mg/m² cont. inf. 46h all on day 1, Repeated every 2 weeks.
  Treatment will be administered until progression, patients' withdrawal of consent, unacceptable toxicity.
  Interventions: Drug: Irinotecan; Drug: Oxaliplatin; Drug: Levoleucovorin; Drug: 5-FU

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 165 mg/m² 1-hour IV day 1
  Other Names: CPT11; Camptosar
Drug: Oxaliplatin — oxaliplatin 85 mg/m² 2-hours IV day 1
  Other Names: L-OHP; Eloxatin
Drug: Levoleucovorin — Levoleucovorin 200 mg/m² 2-hours IV day 1
  Other Names: Fusilev; l-LV
Drug: 5-FU — 5-FU 2800 mg/m² 46-hours flat continuous infusion IV
  Other Names: 5-Fluorouracil
Drug: GM-CSF — GM-CSF 150ug s.c. d3-7 , Repeated every 4 weeks.
  Other Names: Granulocyte Macrophage Colony Stimulating Factor
  Arms: FOLFOXIGIL
Drug: IL-2 — Interleukin-2 100MIU s.c. d8-14 and d17-d28, Repeated every 4 weeks.
  Other Names: Interleukin-2
  Arms: FOLFOXIGIL

SUMMARY:
A randomized phase II trial of FOLFOXIRI in Combination With GM-CSF and IL-2 (FOLFOXIGIL) Versus FOLFOXIRI as First-line Treatment for Patients With Metastatic Colorectal Cancer.

DETAILED DESCRIPTION:
The triple drug regimen FOLFOXIRI (irinotecan, oxaliplatin, fluorouracil, and folinate) for the first-line treatment of metastatic colorectal cancer has shown a significant increase in response rate and overall survival compared to FOLFIRI and FOLFOX. The combination of GOLF chemotherapy with GM-CSF and IL-2（GOLFIG regimen） has shown more active than the standard FOLFOX chemotherapy in first-line mCRC patients，through the chemoimmunomodulatory effects. SO the FOLFOXIGIL chemoimmunotherapy regimen was designed with the same principle to evaluate the antitumor frontline efficacy in comparison with the FOLFOXIRI regimen as first-line treatment of mCRC patients. This is a multicenter, randomized controlled, double-blind, phase II trial.

ELIGIBILITY:
Inclusion Criteria:

* histological or cytological documentation of adenocarcinoma of the colon or rectum.
* unresectable metastatic disease
* age 18 to 75 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or lower if age 70 years or younger or ECOG performance status of 0 if age 71 to 75 years
* at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria measured within 4 weeks prior to registration.
* no previous chemotherapy or target therapy for metastatic disease (adjuvant chemotherapy for non-metastatic disease is allowed if terminated more than 6 months ago).
* adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment:

  * Leukocytes ≥ 3.0 x109/ L, absolute neutrophil count (ANC) ≥ 1.5 x109/ L, platelet count ≥ 100 x109/ L, hemoglobin (Hb) ≥9g/ dL.
  * Total bilirubin ≤ 1.5 x the upper limit of normal (ULN).
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x ULN.
  * Alkaline phosphatase limit ≤ 5x ULN.
  * Amylase and lipase ≤ 1.5 x the ULN.
  * Serum creatinine ≤ 1.5 x the ULN.
  * Calculated creatinine clearance or 24 hour creatinine clearance ≥ 50 mL/ min.

Exclusion Criteria:

* previous palliative chemotherapy for metastatic disease
* previous chemotherapy including irinotecan or oxaliplatin
* symptomatic cardiac disease, myocardial infarction in the last 24 months or uncontrolled arrhythmia
* active infections
* pregnancy or lactation at the time of study entry.
* inflammatory bowel disease
* major autoimmune diseases
* acquired immunosuppression (AIDS or major immunosuppressive agents)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-20 (Estimated); Primary Completion 2019-07-20 (Estimated); Study Completion 2020-07-20 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate at 10 months | PFS rate at 10 months from study entry
  PFS by investigator-reported measurements according to CT image. PFS was calculated from the day of randomization to the date of first documented progression disease (PD) , or death from any cause.
  PD was defined as Overall Response by RECIST criteria v1.1 according to CT image.

SECONDARY OUTCOMES:
Response rate | up to 12 months
  CR + PR rate according to the RECIST version 1.1 guidelines.
Toxicity | up to 12 months
  Toxicity assessed using the NCI common toxicity criteria, version 4.01
Overall survival time | Up to 30 months
  OS was calculated from the date of randomization to death from any cause.
Progression free survival | Up to 18 months
  PFS was calculated from the day of randomization to the date of first documented progression, or death from any cause.
Quality of life (QLQ C30) | Quality of life was evaluated every 2 weeks during treatment and every 8 weeks during follow up (36 months)
  Scores according to EORTC QLQ-C30 scoring manual

CONTACTS AND LOCATIONS:
Overall Officials: Rongbo Lin, MD, Study Chair — Fujian Cancer Hospital
Locations (1):
- Rongbo Lin, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No